CLINICAL TRIAL: NCT01525394
Title: A Double-Blind Study in Healthy Volunteers to Assess the Effect of E7080 on the QTc Interval
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: E7080-A001-002
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2012-04

CONDITIONS: Refractory Solid Tumors; Lymphomas
Keywords: lymphomas; Refractory solid tumors
MeSH Terms: conditions — Lymphoma | interventions — lenvatinib; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Lenvatinib Capsules (Experimental)
  Interventions: Drug: Lenvatinib
- Moxifloxacin tablets (Active Comparator)
  Interventions: Drug: Moxifloxacin 400 mg
- Placebos (Placebo Comparator)
  Interventions: Drug: Placebos (matched to 4 mg and 10 mg lenvatinib capsules).

INTERVENTIONS:
Drug: Lenvatinib — 32 mg will be administered orally as three 4 mg and two 10 mg capsules as a single dose.
  Other Names: E7080
  Arms: Lenvatinib Capsules
Drug: Moxifloxacin 400 mg — Moxifloxacin 400 mg will be administered orally as one 400 mg tablet.
  Arms: Moxifloxacin tablets
Drug: Placebos (matched to 4 mg and 10 mg lenvatinib capsules). — The Placebo dose will consist of three 4 mg and two 10 mg placebo capsules.
  Arms: Placebos

SUMMARY:
This is a double-blind (vis-a-vis lenvatinib), randomized, placebo-controlled, three-treatment, three-way crossover study in healthy subjects. There are two phases in this study: Pre-Randomization and Randomization. The Pre-Randomization Phase consists of Screening and Baseline Period 1. The Randomization Phase consists of five periods: Treatment Period 1, Baseline Period 2, Treatment Period 2, Baseline Period 3, and Treatment Period 3. Completion of study termination procedures will be performed at Visit 11.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be included in this study:

1. Normal, healthy male and female subjects greater than or equal to 18 years of age at the time of informed consent.
2. All females must have a negative serum human chorionic gonadotropin (hCG) pregnancy test result at Screening and Baseline. Females of child-bearing potential must agree to use a medically acceptable method of contraception (e.g., abstinence, an intrauterine device (IUD), a double-barrier method such as condom + spermicide or condom + diaphragm with spermicide, a contraceptive implant, an oral contraceptive or have a vasectomized partner) throughout the entire study period and for 30 days after study drug discontinuation. The only subjects who will be exempt from this requirement are postmenopausal women (defined as greater than age 50 and at least 12 months of amenorrhea) or subjects who have been sterilized surgically or who are otherwise proven sterile (e.g., bilateral tubal ligation with surgery at least 6 months prior to dosing, hysterectomy, or bilateral oophorectomy with surgery at least 2 months prior to dosing). All women who are of reproductive potential and who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 12 weeks prior to dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.
3. Male patients who are not abstinent or have undergone a successful vasectomy, who are partners of women of childbearing potential must use, or their partners must use a highly affective method of contraception (e.g., condom + spermicide, condom + diaphragm with spermicide, IUD) starting for at least one menstrual cycle prior to starting study drug(s) and throughout the entire study period and for 30 days (longer if appropriate) after the last dose of study drug. Those with partners using hormonal contraceptives must also be using an additional approved method of contraception (as described previously).
4. Partners of male and female subjects must use an effective method of contraception (e.g., barrier method, IUD), commencing prior to or at initiation of study drug and continuing for the duration of the study and for 30 days after study drug discontinuation. All females who are of reproductive potential and who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 12 weeks prior to dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.
5. Voluntarily provide written informed consent prior to any study procedures.
6. Are willing and able to comply with all aspects of the protocol for the duration of the study.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participation in the study:

1. Subjects with any clinically significant abnormality, including a QTc interval of greater than 450 msec, on 12-lead ECG at the time of the Screening Period, Baseline Periods, or 30 minutes before administration of study drug.
2. A history of myocardial infarction, syncope or cardiac arrhythmias.
3. A history of uncontrolled hypertension, defined as a systolic pressure of greater than 140 mm Hg and diastolic pressure of greater than 90 mm Hg.
4. A history of unstable heart disease or additional risk factors for Torsades de Pointes (TdP) including heart failure, hypokalemia, or a family history of congenital long QT syndrome or unexplained cardiac arrest.
5. Subjects with a history of gastrointestinal surgery (hepatectomy, nephrotomy, digestive organ resection, etc.) that may affect PK profiles of lenvatinib.
6. Known intolerance to the study drug or moxifloxacin (Avelox) (or any of the excipients).
7. A positive result from human immunodeficiency virus (HIV), hepatitis A antibody (HAVAb), hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCVAb) tests at Screening.
8. A known or suspected history of drug or alcohol misuse within 6 months prior to Screening, or who have a positive urine drug test or breath alcohol test at Screening.
9. Subjects who participated in another clinical trial of an investigational drug or device within 4 weeks prior to dosing.
10. Subjects who received blood products within 4 weeks, or donated blood within 8 weeks, or donated plasma within one week of dosing.
11. Subjects who have engaged in heavy exercise within 2 weeks prior to check-in (e.g., marathon runners, weight lifters, etc.).
12. Females who are pregnant or breastfeeding.
13. Subjects who are unwilling or unable to abide by the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the potential for QT/QTc prolongation by 32 mg lenvatinib using a placebo control and moxifloxacin as the positive control. | 2 months

SECONDARY OUTCOMES:
To evaluate the safety of lenvatinib in healthy subjects. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Shumaker, Study Director — Eisai Inc.
Locations (1):
- Charles River, Tacoma, Washington, United States